CLINICAL TRIAL: NCT04040400
Title: A Phase I/II Study of Intraoperative Radiotherapy for Patients With Large Brain Metastases Treated With Neurosurgical Resection
Brief Title: Study of Intraoperative Radiotherapy for Patients With Large Brain Metastases Treated With Neurosurgical Resection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: per DMSC request
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Shiao Yuo Woo,M.D., Principal Investigator, University of Louisville
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19.0619 BCC-IORT-BM
Record Dates: First submitted 2019-07-20; First posted 2019-07-31 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: The resection procedure should be performed with image guidance (neuronavigation) with standard surgical technique.
  Optimal balloon applicator size will be selected with accordance to tumor bed/cavity geometry and adjacent normal brain parenchyma by the team of surgeons and radiation oncologists.
  The radiation oncologist will place the miniature x-ray source inside the balloon shaped catheter placed inside the tumor cavity. Radiotherapy will be initiated by the treating radiation oncologist for a defined time interval calculated by the machine planning software.
  After IORT has been delivered, the surgeon will remove the balloon applicator. Surgery will be continued in the regular fashion without additional requirements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment Arm (Experimental): intraoperative radiotherapy (IORT) arm
  Interventions: Radiation: intraoperative radiotherapy (IORT)

INTERVENTIONS:
Radiation: intraoperative radiotherapy (IORT) — intraoperative radiotherapy (IORT) during brain tumor resection to establish a maximum tolerated dose (MTD) through a dose-escalation trial using intraoperative radiotherapy (IORT)

SUMMARY:
The primary purpose of this study is to establish a maximum tolerated dose (MTD) through a dose-escalation trial using intraoperative radiotherapy (IORT) following neurosurgical resection for large brain metastases, and to determine the progression-free survival rate as in the recurrence rate of treated brain metastasis.

DETAILED DESCRIPTION:
The potential for delivering ablative doses of radiation to the tumor bed while simultaneously sparing normal brain parenchyma from significant doses of radiation and reducing the potential for tumor repopulation has led to interest in the use of intraoperative radiotherapy (IORT) for brain metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be ≥ 18 years of age.
2. Participants must have a Karnosfky performance status of ≥ 50%.
3. Participants must not have had prior intracranial radiation.
4. Participants must have a life expectancy greater than 3 months.
5. Participants must have a preoperative MRI Brain T1-Gadolinum enhanced scan demonstrating a non-dural based lesion with greatest diameter ≥ 2.5 cm.
6. Sufficient distance (≥ 2cm) of the intracranial lesion from optic structures (optic chiasm and bilateral optic nerves) and brainstem to meet established normal structure dose limits.
7. Subject or subject's legal representative to provide signed/written informed consent to participate in the study protocol.
8. Surface of balloon applicator must be ≥ 1cm from skin overlying closest portion of calvarium.
9. Participants may remain on systemic therapy if they are receiving immunotherapy (anti-PD1, anti-PDL1, anti-CTLA-4), capecitabine, temozolomide, etoposide, vinorelbine, pemetrexed, lapatinib, traztuzumab, bevacizumab, mTor or ALK targeted agents with no break prior to initiating IORT.

9.1 Participants receiving cisplatin, methotrexate, taxanes, tyrosine kinase inhibitors, or BRAF targeted agents must have a seven day washout period prior to receiving IORT.

9.2 Participants receiving doxorubicin, T-DM1, or antibody-drug conjugates must have a fourteen day washout period prior to receiving IORT.

9.3. Participants receiving all other concurrent systemic agents will undergo consideration for a washout period prior to receiving IORT at the discretion of the study principal investigator.

Exclusion Criteria:

1. Participants may not be pregnant or breast-feeding.
2. Patients must not have dural lesions or leptomeningeal disease.
3. Patients must not have psychiatric or social conditions limiting adherence to protocol guidelines.
4. Patients must not have contraindications to anesthesia, surgery, or MR imaging with Gadolinium injection.
5. Patients must not have a frozen section diagnosis of small cell carcinoma, lymphoma, germinoma or non-malignant histology.
6. Patients with additional unresected brain metastases must have a limited number of lesions/or volume of intracranial disease amenable to stereotactic radiotherapy at the discretion of the study principal investigator.
7. Patients deemed to require postoperative whole brain radiotherapy should be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaio Woo, MD, Principal Investigator — University of Louisville, JGBrown Cancer Center
Locations (1):
- University of Louisville, James Graham Brown Cancer Center, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share individual participant data with other researchers outside of this clinical trial's investigation team

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm Intraoperative Radiotherapy (IORT): Cohort 1 received 18 Gy. Intraoperative radiotherapy (IORT) during brain tumor resection.
- Cohort 2: Planned dose: 21 Gy. No patient accrued in this cohort.
- Cohort 3: Planned dosage 24 Gy. No patient accrued in this cohort.
Period: Cohort 1
Arm/Group | Treatment Arm Intraoperative Radiotherapy (IORT) | Cohort 2 | Cohort 3
Started | 5 | 0 | 0
Completed | 5 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Cohort 1:
Arm/Group | Treatment Arm Intraoperative Radiotherapy (IORT) | Cohort 2 | Cohort 3
Started | 5 | 0 | 0
Completed (1 participant died of respiratory failure unrelated to treatment.) | 4 | 0 | 0
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intraoperative Radiotherapy Treatment Arm: Participants receiving Intraoperative Radiotherapy with Neurosurgical Resection.
Arm/Group | Intraoperative Radiotherapy Treatment Arm
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants] — Population: 3 screen failed and 1 withdrew and were unable to be analyzed.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 2
    >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 3 screen failed and 1 withdrew and were not analyzed.
  Participants
    Female | 1
    Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Established Maximum Tolerated Dose
Description: Maximum tolerated dose will be determined by classical 3+3 dose-escalation design. Toxicity will be measured using the National Cancer Institute Common terminology criteria for adverse events (version 5.0).
  The first dose of 18Gy will be administered to the first 3 subjects, after 90 days from treatment a safety assessment for dose limiting toxicities will be done to determine if the next 3 subject will escalation to dose of 21Gy or receive 18Gy.
  If escalation to 21Gy is permitted, then after 90 days from treatment a safety assessment for dose limiting toxicities will be done to determine if next cohort of 3 subjects will escalate to a dose of 24Gy or receive 21Gy. The highest dose level to be administered will be 24 Gy if permitted by safety assessments.
Time Frame: Phase I cohorts; 90 days from treatments
Measure: Count of Participants; unit: Participants
Groups:
- IORT Treatment Arm: Participants receiving Intraoperative Radiotherapy with Neurosurgical Resection.
Arm/Group | IORT Treatment Arm
Number analyzed (Participants) | 5
Participants
  18 Gy | 5
  21 Gy | 0
  24 Gy | 0

2. Primary Outcome: Number of Participants With Adverse Events
Description: Number of adverse events reported per participant.
Time Frame: 12 months
Population: participants that received intraoperative radiation.
Measure: Number; unit: participants
Arm/Group | IORT Treatment Arm
Number analyzed (Participants) | 5
participants | 5

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected from date of first patient enrollment to close of study due to all participant death/loss to follow-up, a period of 2 years from study activation.
Description: Zero participants accrued in cohorts 2 and 3.
Groups:
- Cohort 1: 18 Gy: Participants receiving Intraoperative Radiotherapy with Neurosurgical Resection.
- Cohort 2: 21 Gy; Cohort 3: 24 Gy: Planned participants receiving Intraoperative Radiotherapy with Neurosurgical Resection.
Arm/Group | Cohort 1: 18 Gy | Cohort 2: 21 Gy | Cohort 3: 24 Gy
All-Cause Mortality (participants affected / at risk) | 4/5 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 5/5 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/5 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 18 Gy (N=5) | Cohort 2: 21 Gy (N=0) | Cohort 3: 24 Gy (N=0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA — AE Grade 4
Acute Kidney Injufy (Renal and urinary disorders) | 1 (1) | NA | NA — AE Grade 3
Worsening Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA | NA — AE Grade 3 The tumor was removed prior to the XOFT treatment and patient later admitted on for recurrence. Same site, left occipatal brain mass.
Thromboembolic Event (Blood and lymphatic system disorders) | 1 (1) | NA | NA — AE Grade 3
Meningitis - Bacterial (Infections and infestations) | 1 (1) | NA | NA — AE Grade 3
Altered Mental Status (Nervous system disorders) | 1 (1) | NA | NA — AE Grade 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 18 Gy (N=5) | Cohort 2: 21 Gy (N=0) | Cohort 3: 24 Gy (N=0)
XOft Overdose (General disorders) | 1 (1) | NA | NA — Deviation: Patient was accidentally given 24 Gy at first dose due to calculation error. No additional adverse event found to be related to overdose.
Worsening Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA | NA — AE Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT04040400/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT04040400/ICF_001.pdf